CLINICAL TRIAL: NCT06098495
Title: Looking for a Blood Epigenetic Signature to Predict Female Infertility
Acronym: FIB_CARIPLO
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Valeria Stella Vanni, Doctor, Università Vita-Salute San Raffaele
Other Study IDs: FIB_CARIPLO_1.0
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, Oocyte granulosa cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- infertile women (unexplained, tubal, mild male factor): women belonging to couples selected for homologous IVF due to an unexplained, tubal or mild male factor
- fertile women: women without any infertility history who are attempting to conceive naturally
  Interventions: Genetic: search for epigenetic profile of infertility
- infertile women (ovarian factor): women selected for homologous IVF for different reason og chohort 1
  Interventions: Genetic: search for epigenetic profile of infertility
- recurrent pregnancy loss: women affected by idiopathic recurrent pregnancy loss
  Interventions: Genetic: search for epigenetic profile of infertility

INTERVENTIONS:
Genetic: search for epigenetic profile of infertility — examine the epigenetic profile of DNA extracted from MGCs and blood sample
  Groups: fertile women; infertile women (ovarian factor); recurrent pregnancy loss

SUMMARY:
The present research project aims to study the DNAm mechanisms underlying the reduction of fertility due to the progressive depletion of oocyte quality. Specifically, our project aims to build an epigenetic clock for MGCs by using outcomes that are certainly related to female fertility. The validation of such findings will be carried out on peripheral blood in order to guarantee its non-invasiveness and allow for any clinical transferability. In order to identify a blood epigenetic signature able to predict female infertility, we planned to explore the problem from different points of view by conducting several studies in different settings.

ELIGIBILITY:
Inclusion Criteria:

* 18< age <43, Infertile woman undergoing ART, recurrent pregnancy loss

Exclusion Criteria:

* age < 18 or > 44, previous ovarian surgery, severe male factor infertility

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: Infertile woman undergoing ART, women affected by recurrent pregnancy loss, women attempting to conceive naturally
Sampling Method: Non-Probability Sample
Enrollment: 1456 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
differences of DNA methylation in granulosa cells of patients undergoing ART | 3 years
  The epigenetic profile of DNA extracted from granulosa cells of patients undergoing ART (COHORT1) will be examined to identify position and region's differences of DNA methylation in pregnant women (fertile women) and in who does not get pregnant (infertile women)
differences of DNA methylationin the peripheral venous blood of patients undergoing ART | 3 years
  search for this methylation difference found in the granulosa cell sample, also in the peripheral venous blood of these same patients
differences of DNA methylationin the peripheral venous blood of women attempting to conceive naturally | 3 years
  The specific epigenetic modification will be searched in the peripheral venous blood of women attempting to conceive naturally (COHORT2)
differences of DNA methylationin the peripheral venous blood of new patients undergoing ART | 3 years
  The specific epigenetic modification will be searched in the peripheral venous blood of two new cohorts of patients referred to PMA centres.
impact of exogenous pro-inflammatory factors | 3 years
  on all the above cohorts will be investigated, via online questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita Salute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
publication of the results at the end of the trial